CLINICAL TRIAL: NCT00570505
Title: Effectiveness and Safety Study of LAP-BAND Treatment in Subjects With BMI >/= 30 kg/m2 and < 40 kg/m2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Apollo Endosurgery, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LBMI-001
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Results first posted 2012-12-03 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LapBand (Experimental): All subjects who receive the LAP-BAND System.
  Interventions: Device: LAP-BAND System

INTERVENTIONS:
Device: LAP-BAND System — Reduction of food intake due to creation of smaller stomach pouch

SUMMARY:
The purpose of this study is to determine whether the LAP-BAND system is safe and effective in subjects with BMI ≥ 30 kg/m2 and < 40 kg/m2.

DETAILED DESCRIPTION:
LBMI-001 is a multi-center, prospective, longitudinal, non-randomized study whose purpose is to determine whether the LAP-BAND system is safe and effective in subjects with BMI ≥ 30 kg/m2 and < 40 kg/m2. Primary and secondary outcome measures were analyzed at 1 year post LAP-BAND implantation. Subjects continued to be followed for 5 years post-implantation, and 5 year data was evaluated in Post-Hoc outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Have a BMI ≥ 30 kg/m2 and < 35 kg/m2 (with or without comorbid conditions) or a BMI ≥ 35 kg/m2 and < 40 kg/m2 without severe comorbid conditions
* Have a history of obesity for at least 2 years and have failed more conservative weight-reduction alternatives, such as supervised diet, exercise and behavior modification programs

Exclusion Criteria:

* Subject history of congenital or acquired anomalies of the gastrointestinal tract
* Severe cardiopulmonary or other serious or uncontrolled organic disease
* Severe coagulopathy; hepatic insufficiency or cirrhosis
* History of bariatric; gastric; or esophageal surgery
* History of intestinal obstruction or adhesive peritonitis
* History of esophageal dysmotility disorders
* Type I diabetes

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2007-11; Primary Completion 2009-10 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle, Washington, United States

REFERENCES:
- [Result] Michaelson R, Murphy DK, Gross TM, Whitcup SM; LAP-BAND Lower BMI Study Group. LAP-BAND for lower BMI: 2-year results from the multicenter pivotal study. Obesity (Silver Spring). 2013 Jun;21(6):1148-58. doi: 10.1002/oby.20477. PMID 23637029

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 155 Subjects were enrolled per protocol (defined as signing the informed consent). After enrollment, 4 subjects withdrew consent prior to treatment, and 2 subjects were not implanted due to ineligibility discovered during screening. This resulted in 149 subjects starting the study and receiving treatment with the LAP-BAND System.
Period: Overall Study
Arm/Group | LapBand
Started | 149
Completed | 108 (The number of subjects completing the 60-month study)
Not Completed | 41
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 23
Not completed — Other loss to follow-up | 4

BASELINE CHARACTERISTICS:
Groups:
- LapBand: Subjects implanted with the LapBand(R) Adjustable Gastric Band System
Arm/Group | LapBand
Number analyzed (Participants) | 149
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 147
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.28 (9.304)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 149

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects Attaining Clinically Successful Weight Loss ( ≥ 30% EWL) at 1 Year Post LAP-BAND Implantation
Description: The percent of subjects attaining clinically successful weight loss at 1 year post LAP-BAND implantation. Clinically successful weight loss was defined as ≥ 30% Excess Weight Loss (%EWL), where %EWL was weight loss divided by excess weight multiplied by 100.
Time Frame: One year
Population: Intent-to-treat (ITT)
Measure: Number; unit: percentage of subjects
Arm/Group | LapBand
Number analyzed (Participants) | 143
percentage of subjects | 83.9

2. Secondary Outcome: Percent Weight Loss
Description: Percent weight loss was defined as weight loss divided by baseline weight, multiplied by 100. Weight loss was equal to baseline weight minus the follow-up visit weight. Excess weight = baseline weight minus ideal weight, where ideal weight was determined based on a BMI of 25 kg/m2.
Time Frame: Baseline through 12 months
Population: Intent-to-treat (ITT)
Measure: Mean (Standard Deviation); unit: percentage of weight loss
Arm/Group | LapBand
Number analyzed (Participants) | 143
percentage of weight loss | 18.32 (8.516)

3. Secondary Outcome: Change in Comorbid Conditions Related to Obesity
Description: Percent of subjects whose baseline comorbid condition of Type 2 diabetes, dyslipidemia, and hypertension resolved (i.e., was rated as "none" on a severity scale of none, mild, moderate, or severe) 12 months after implantation.
Time Frame: 12 months
Population: Subjects who had the specific comorbid condition at baseline (Diabetes n = 6, Dyslipidemia n = 29, Hypertension n = 27)
Measure: Number; unit: percentage of subjects
Arm/Group | LapBand
Number analyzed (Participants) | 143
percentage of subjects
  Diabetes Type II (n = 6) | 33.3
  Dyslipidemia (n = 29) | 27.6
  Hypertension (n = 27) | 22.2

4. Secondary Outcome: Change in Quality of Life
Description: Change in quality of life was assessed using the Impact of Weight on Quality of Life-Lite (IWQOL-Lite) Total Score, which ranges from 0 (worst) to 100 (best). The mean change from baseline to 12 months in IWQOL-Lite Total Score is reported.
Time Frame: 12 months
Population: Intent-to-treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LapBand
Number analyzed (Participants) | 143
units on a scale | 28.03 (17.274)

5. Post Hoc Outcome: Percent of Subjects Attaining Clinically Successful Weight Loss ( ≥ 30% EWL) at 5 Years Post LAP-BAND Implantation
Description: The percent of subjects who attained clinically successful weight loss (ie, ≥ 30% Excess Weight Loss) at year 5 post LAP-BAND implantation. Percent EWL =(weight loss divided by excess weight)*100. Excess Weight was defined as Baseline Weight - Ideal Weight, where Ideal Weight was a BMI of 25 kg/m2.
Time Frame: 5 years
Population: Intent-to-treat (ITT)
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | LapBand
Number analyzed (Participants) | 108
percentage of subjects | 76.9 [67.75 to 84.43]

6. Post Hoc Outcome: Subject Percent Excess Weight Loss (5 Years)
Description: The mean percent excess weight loss (%EWL) for subjects at month 60. Percent EWL = (weight loss divided by excess weight)*100.
Time Frame: 5 years
Population: Intent-to-treat (ITT)
Measure: Mean (Standard Deviation); unit: percentage of excess weight loss
Arm/Group | LapBand
Number analyzed (Participants) | 108
percentage of excess weight loss | 62.74 (41.131)

7. Post Hoc Outcome: Change in Obesity Related Comorbid Conditions (5 Years)
Description: Percent of subjects whose baseline comorbid condition of Type 2 diabetes, dyslipidemia, and hypertension resolved 5 years post LAP-BAND implantation. Diabetes resolution was defined as HbA1c ≤ 6% and no diabetes medication usage. Dyslipidemia resolution was defined as HDL ≥ 60 mg/dL, LDL < 100 mg/dL, triglycerides < 150 mg/dL, and total cholesterol < 200 mg/dL. Hypertension resolution was defined as systolic blood pressure < 140 mm Hg.
Time Frame: 5 years
Population: Subjects who had the specific comorbid condition at screening (Type 2 Diabetes n=5, Dyslipidemia n=45, Hypertension n=49)
Measure: Number; unit: percentage of subjects
Arm/Group | LapBand
Number analyzed (Participants) | 108
percentage of subjects
  Type 2 Diabetes (n=5) | 40.0
  Dyslipidemia (n=45) | 4.4
  Hypertension (n=49) | 12.2

8. Post Hoc Outcome: Change in Quality of Life (5 Years)
Description: Change in quality of life was assessed using the Impact of Weight on Quality of Life-Lite (IWQOL-Lite) Total Score, which ranges from 0 (worst) to 100 (best). The mean change from baseline to 5 years in IWQOL-Lite Total Score is reported.
Time Frame: 5 years
Population: Intent-to-treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LapBand
Number analyzed (Participants) | 104
units on a scale | 29.23 (19.397)

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | LapBand
Serious Adverse Events (participants affected / at risk) | 18/149
Other Adverse Events (participants affected / at risk) | 145/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LapBand (N=149)
Abdominal cavity abscess (Gastrointestinal disorders) | 1 (1)
Band erosion (Gastrointestinal disorders) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Dysphagia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastric outlet obstruction (Gastrointestinal disorders) | 5 (5)
Esophageal spasms (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastric prolapse (Gastrointestinal disorders) | 4 (4)
Umbilical hernia contained LAP-BAND tubing (General disorders) | 1 (1)
Recurrent gastric stricture (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Band slip (Gastrointestinal disorders) | 4 (6)
Hiatal hernia (Gastrointestinal disorders) | 1 (1)
Biliary colic (Renal and urinary disorders) | 1 (1)
Cholelithiasis (Renal and urinary disorders) | 1 (1)
Pouch dilation (Gastrointestinal disorders) | 1 (1)
Esophageal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LapBand (N=149)
Vomiting (Gastrointestinal disorders) | 104 (104)
Dysphagia (Gastrointestinal disorders) | 73 (73)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 77 (77)
Dyspepsia (Gastrointestinal disorders) | 30 (30)
Nausea (Gastrointestinal disorders) | 24 (24)
Gastric dilation (Gastrointestinal disorders) | 19 (19)
Abdominal pain (Gastrointestinal disorders) | 16 (16)
Regurgitation of food (Gastrointestinal disorders) | 16 (16)
Esophageal dilation (Gastrointestinal disorders) | 12 (12)
Abdominal pain upper (Gastrointestinal disorders) | 11 (11)
Constipation (Gastrointestinal disorders) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 8 (8)
Post procedural pain (Injury, poisoning and procedural complications) | 29 (29)
Medical device complication (Injury, poisoning and procedural complications) | 25 (25)
Implant site pain (General disorders) | 12 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Anemia (Blood and lymphatic system disorders) | 8 (8)
Dehydration (Metabolism and nutrition disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 120 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.